CLINICAL TRIAL: NCT05440513
Title: Trans Ureteral Sympathectomy of the Kidney Study Using the Verve Medical Phoenix ™ System
Brief Title: A Study of Non-Vascular Renal Denervation Using the Verve Medical Phoenix ™ System
Acronym: TUSK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Verve Medical, Inc (Industry)
Collaborators: Clinical Accelerator (Industry); Israeli-Georgian Medical Research Clinic Helsicore (Unknown); Pineo Medical Ecosystem (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0002
Record Dates: First submitted 2022-06-23; First posted 2022-07-01 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Renal Pelvic Denervation (Experimental): Using the natural orifice of the urethra, the ureters are accessed (bilaterally and in sequence), to allow for an ablation device to be placed into the renal pelvis where RF energy is delivered to ablate renal nerves.
  Interventions: Device: Renal Pelvic Denervation (bilateral)

INTERVENTIONS:
Device: Renal Pelvic Denervation (bilateral) — Using the natural orifice of the urethra, the ureters are accessed (bilaterally and in sequence), to allow for an ablation device to be placed into the renal pelvis where RF energy is delivered to ablate renal nerves.
  Other Names: renal nerve ablation; renal sympathectomy

SUMMARY:
The aim of the study is to assess the safety and effectiveness of a novel device for renal denervation to lower blood pressure in people with uncontrolled hypertension. Prior studies demonstrate the potential benefit of renal denervation in hypertension, though these studies primarily denervate the kidneys by passing catheters through the arteries in the groin into the renal arteries. The TUSK study utilizes the Phoenix system to perform denervation by advancing the device (a thin electrode) through the urinary tract into the kidneys where radiofrequency energy is briefly applied to denervate the kidneys.

DETAILED DESCRIPTION:
Up to 20 patients with uncontrolled hypertension will be treated with the PhoenixTM renal pelvic denervation system, whether or not receiving background medical therapy.

Qualification will be based on documented uncontrolled hypertension by 24-hour ambulatory blood pressure monitoring. Those qualifying will be expected to maintain their medical therapy without changes until after the primary effectiveness assessment two months later.

Following baseline testing, patients will undergo renal pelvic denervation under anesthesia and remain in the hospital overnight. The denervation device is inserted through the urethra into each kidney and all devices are removed at the completion of the procedure. Radiofrequency energy is administered for a single 2-minute treatment period in each kidney.

Follow up visits will extend to one year. Patients will complete medication logs along with repeat assessment of blood pressure in office and via 24-hour ambulatory blood pressure monitor. Follow up testing will also include imaging studies of the kidneys.

ELIGIBILITY:
Key Inclusion Criteria:

* Off-med group: (1) Ambulatory mean daytime SBP ≥140 mmHg in patients never treated for hypertension or after being taken off anti-hypertension medications for 4 weeks before ambulatory blood pressure assessment. (2) Ambulatory daytime SBP and DBP less than 170/105 mmHg. (3) Subjects will not be on ANY anti-hypertension medications or will be willing to discontinue current anti-hypertension medications.
* On-med group: (1) Subjects who are currently taking 1, 2, or 3 anti-hypertensive medications. (2) Ambulatory mean daytime SBP ≥135 mmHg. (3) Ambulatory daytime SBP and DBP less than 170/105 mmHg.

Exclusion Criteria:

* Females who are either pregnant or breastfeeding.
* Office SBP or DBP ≥180/110 mmHg.
* Untreated urinary tract infection.
* Renal collecting system is compromised, and subject cannot undergo routine cystoscopy and retrograde pyelogram.
* Dialysis patients.
* Renal transplant patients.
* Subjects on the following medications, clonidine, guanfacine and methyldopa.
* Known secondary causes of hypertension such as adrenal disease, renal artery stenosis, renovascular hypertension.
* Subjects with glomerulonephritis or interstitial nephritis or eGFR < 45 ml/min/1.73m2.
* Type I diabetes mellitus.
* Stenotic valvular heart disease for which reduction of blood pressure would be hazardous.
* Subjects with orthostatic hypotension.
* Myocardial infarction, unstable angina, or stroke in the prior 6 months.
* Any medical condition (including psychiatric disease) that would interfere with conducting the study or would not be in the best interest of the subject.
* Inability of the subject to provide informed consent.
* Subjects with sleep apnea.
* Patients taking any drugs that affect blood pressure through off target effects
* Patients with any clinical condition that can affect blood pressure or require the use of drugs that can affect blood pressure. e.g. NSAIDs, steroids, cold remedies.
* Patients who may require any procedure that can affect blood pressure.
* Patients who work a night shift.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in mean daytime systolic blood pressure | Month 2
  Mean daytime systolic blood pressure determined from ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Change in mean 24-hour systolic blood pressure | Month 2
  Mean 24-hour systolic blood pressure determined from ambulatory blood pressure monitoring
Change in automated office systolic blood pressure | Month 2
  Automated office blood pressure measured after resting and in triplicate
Safety of renal pelvic denervation | Month 2
  Number of subjects with serious adverse events, treatment-emergent adverse events and adverse events assessed, including evidence for acute kidney injury and hypertension-related morbidity

OTHER OUTCOMES:
Effect on renal function | Month 2
  Effects on serum creatinine
Effect on index of renal function | Month 2
  Effects on estimated glomerular filtration rate
Effects on ABPM at month 6 (durability of effects) | Through month 6
  ABPM performed during follow-up
Effects on ABPM month 12 (durability of effects) | Through month 12
  ABPM performed during follow-up
Effects on OBM at month 6 (durability of effects) | Through month 6
  OBP performed during follow-up
Effects on OBP at month 12 (durability of effects) | Through month 12
  OBP performed during follow-up
Safety of renal pelvic denervation | Through month 6
  Number of subjects with serious adverse events, treatment-emergent adverse events and adverse events assessed, including evidence of acute kidney injury
Safety of renal pelvic denervation | Through month 12
  Number of subjects with serious adverse events, treatment-emergent adverse events and adverse events assessed, including evidence of acute kidney injury

CONTACTS AND LOCATIONS:
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hering D, Hubbard BS, Weber MA, Heuser RR. Impact of Renal Pelvic Denervation on Systemic Hemodynamics and Neurohumoral Changes in a Porcine Model. Am J Nephrol. 2021;52(5):429-434. doi: 10.1159/000516186. Epub 2021 May 26. PMID 34038910
- [Derived] Hering D, Nikoleishvili D, Imedadze A, Dughashvili G, Klimiashvili Z, Bekaia E, Shengelia T, Kobalava M, Goguadze O, Emukhvari T, Druker V, Sackner-Bernstein J, Weber MA. Transurethral Renal Pelvic Denervation: A Feasibility Trial in Patients with Uncontrolled Hypertension. Hypertension. 2022 Dec;79(12):2787-2795. doi: 10.1161/HYPERTENSIONAHA.122.20048. Epub 2022 Oct 18. PMID 36254733